CLINICAL TRIAL: NCT01130363
Title: Determination of a Possible Association of Fundic Gland Polyps With the Use of Proton Pump Inhibitor Drugs
Brief Title: Fundic Gland Polyps and Proton Pump Inhibitor (PPI) Drugs
Status: Terminated | Type: Observational
Why Stopped: Poor Enrollment
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAC2805
Record Dates: First submitted 2010-05-21; First posted 2010-05-26 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Fundic Gland Polyps
Keywords: Proton Pump Inhibitor; Gastric carcinoid tumors; Gastric cancer; Fundic Gland Polyps
MeSH Terms: conditions — Polyposis, Gastric; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw: A fasting serum gastrin (FSG) level will be obtained to evaluate for hypergastrinemia at a follow-up visit after EGD. Approximately 4 cc's of blood is required. As many patients have been on long term PPI therapy, the FSG level is one method of determining whether the patient is on super-therapeutic levels of PPI which may need to be adjusted.
  Biopsy specimens: Gastric fundic gland polyps found during endoscopy will have biopsies taken of the polyp, adjacent normal gastric body or fundus, and from the antrum.
  Histological evaluation of biopsy specimens: Biopsies will be stained with H&E as well as neuroendocrine cell markers to assess for the presence of ECL cell hyperplasia. Paraffin-fixed tissue will be stored for future biological analysis. This will only be done after all clinically relevant analyses are completed and only if adequate tissue remains.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Fundic Gland Polyps on PPI: Patients found to have fundic gland polyps on endoscopic evaluation that have also been prescribed and regularly take a proton pump inhibitor.
- Fundic Gland Polyp not on PPI: Patients found to have fundic gland polyps on endoscopic evaluation that have not been prescribed a proton pump inhibitor.
- Group 3 (Control Group): Individuals who are prescribed proton pump inhibitor but are not found to have fundic gland polyps on endoscopic evaluation.

SUMMARY:
The class of proton pump inhibitor (PPI) medications such as omeprazole has proven extremely effective in the treatment and prevention of gastric and duodenal ulcers. Although the FDA approval for PPI therapy is limited to 6-8 weeks, many individuals remain on these agents for years, and human studies have suggested that long-term use of a PPI can result in enterochromaffin-like (ECL) cell hyperplasia, as well as being associated with the development of fundic-gland polyps of the stomach. These findings raise the concern of the possibility that long-term use of PPIs may predispose to the development of neuroendocrine tumors in patients. The investigators aim to examine clinical parameters, including history of PPI use and fasting gastrin levels, as well as histologic characteristics (particularly the presence of ECL-cell hyperplasia) of patients found to have fundic gland polyps during endoscopy. The investigators hypothesize that there is a correlation between fundic gland polyps of the stomach and the use of proton pump inhibiter medications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above.
* Able and willing to sign informed consent.
* The patient had a gastric fundic gland polyp detected on EGD that was removed and sent to pathology or patient had no fundic gland polyps on EGD but are on PPIs and will serve as controls.

Exclusion Criteria:

* Unwilling or unable to sign informed consent for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals found to have fundic gland polyps on endoscopic evaluation and are on proton pump inhibitor (PPI), individuals found to have fundic gland polyps on endoscopic evaluation but are not on PPI or patients on PPI but had no fundic gland polyps found on endoscopic evaluation (control group).
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2006-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with fundic gland polyps and PPI use that have a higher gastric pH | Up to 1 year
  We aim to examine clinical parameters, including history of PPI use and fasting gastrin levels, as well as histologic characteristics (particularly the presence of ECL-cell hyperplasia) of patients found to have fundic gland polyps during endoscopy. We believe there is a correlation between fundic gland polyps of the stomach and use of proton pump inhibiter medications.

CONTACTS AND LOCATIONS:
Overall Officials: Harold Frucht, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States